CLINICAL TRIAL: NCT06998602
Title: Student Paramedics' Experiences of Compassion Fatigue: a Phenomenological Mixed-methods Study
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Jonathan Robinson, Ph.D, Senior Lecturer in Research Methods, Teesside University
Other Study IDs: 24118
Record Dates: First submitted 2025-05-20; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Compassion Fatigue; Burnout; Paramedical Professional; Occupational Stress
Keywords: Compassion Fatigue; Burnout; Secondary Traumatic Stress; Paramedic Students; Qualitative Research; ProQOL; Phenomenology
MeSH Terms: conditions — Compassion Fatigue; Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explored how student paramedics experience compassion fatigue - a type of emotional and physical exhaustion that can occur when regularly caring for others in distress. The researchers wanted to understand how student paramedics feel about compassion fatigue, how it affects their work, and what kind of support might help them cope.

To do this, a group of student paramedics were interviewed about their personal experiences and also asked to complete a short questionnaire called the Professional Quality of Life Scale (ProQOL). This questionnaire measured their levels of compassion satisfaction (positive feelings from helping others), burnout (emotional exhaustion), and secondary traumatic stress (stress from exposure to others' trauma).

DETAILED DESCRIPTION:
This was a non-interventional, observational, mixed-methods study that used a phenomenological approach to explore student paramedics' experiences and perceptions of compassion fatigue (CF). The study aimed to identify how CF manifests during training, how it affects clinical practice, and which forms of support students believe would be helpful in preventing or managing CF.

Participants were recruited from the BSc (Hons) Paramedic Practice programme at UK University, using purposive, non-probability sampling. Data collection involved two components:

1. Semi-structured interviews conducted online via Microsoft Teams to explore participants' lived experiences.
2. Completion of the Professional Quality of Life (ProQOL) questionnaire, which measured Compassion Satisfaction, Burnout, and Secondary Traumatic Stress.

Interview transcripts were analysed thematically using Braun and Clarke's six-step framework. The ProQOL data were analysed using descriptive statistics and inferential comparisons using both Frequentist and Bayesian analysis, using JASP software. The target sample size was between 3-10. Seven participants completed the study.

Eligible participants were contacted via email by the designated gatekeeper, the course leader. The email outlined that, as student paramedics who had attended clinical placement as part of their course, they were eligible to take part in the study. The email invited them to read the participant information sheet and contact the primary researcher with any questions. Those interested in participating were asked to get in touch to organise receipt of the informed consent form.

Following initial contact, the primary researcher corresponded with interested participants via email to arrange a suitable date and time for the interview. Depending on participant preference, interviews were conducted either on campus or via Microsoft Teams.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible if they are a current Student Paramedic, studying at target University and have attended clinical placement.

Exclusion Criteria:

* There is no exclusion criteria other than mental capacity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Student paramedics enrolled in the BSc (Hons) Paramedic Practice programme at the target University, a higher education institution located in Middlesbrough, UK. Participants were recruited from across multiple year groups, including apprentices, using purposive sampling.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Themes related to student paramedics' experiences of compassion fatigue | Interviews were completed at a single time point, depending on when the voluntary participant joined the study (between the 19th November 2024 and 13th December 2024).
  Key qualitative themes derived from semi-structured interviews with student paramedics, using Braun and Clarke's six-step thematic analysis framework. Themes will reflect participants' lived experiences, perceptions, and coping mechanisms related to compassion fatigue.

SECONDARY OUTCOMES:
Compassion Satisfaction score (ProQOL) | The questionnaire was completed at a single time point, depending on when the voluntary participant joined the study, post-interview (between the 19th November 2024 and 13th December 2024).
  Self-reported scores on the Compassion Satisfaction subscale of the Professional Quality of Life Scale (ProQOL), version 5, and questions are scored on a scale of 1 to 5, and raw scores range between 10 to 50. Higher scores indicate greater compassion satisfaction, representing a more favourable outcome.
  ProQOL questionnaire, was scored according to the official ProQOL scoring guidelines. The ProQOL is a validated measure with acceptable internal consistency across its subscales, commonly used to assess compassion fatigue and related constructs in healthcare professionals.
  Descriptive statistics (mean and standard deviation) were calculated. If appropriate, to explore potential sex differences, statistical comparisons were conducted using both Frequentist and Bayesian approaches, with analyses performed in JASP software.
Burnout score (ProQOL) | The questionnaire was completed at a single time point, depending on when the voluntary participant joined the study, post-interview (between the 19th November 2024 and 13th December 2024).
  Self-reported scores on the Burnout subscale of the Professional Quality of Life Scale (ProQOL), Version 5 , and questions are scored on a scale of 1 to 5, and raw scores range between 10 to 50. Higher scores indicate higher levels of burnout, representing a less favourable outcome.
  ProQOL questionnaire, was scored according to the official ProQOL scoring guidelines. The ProQOL is a validated measure with acceptable internal consistency across its subscales, commonly used to assess compassion fatigue and related constructs in healthcare professionals.
  Descriptive statistics (mean and standard deviation) were calculated. If appropriate, to explore potential sex differences, statistical comparisons were conducted using both Frequentist and Bayesian approaches, with analyses performed in JASP software.
Secondary Traumatic Stress score (ProQOL) | The questionnaire was completed at a single time point, depending on when the voluntary participant joined the study, post-interview (between the 19th November 2024 and 13th December 2024).
  Self-reported scores on the Secondary Traumatic Stress subscale of the Professional Quality of Life Scale (ProQOL), Version 5, and questions are scored on a scale of 1 to 5, and raw scores range between 10 to 50. Higher scores indicate greater levels of secondary traumatic stress, representing a less favourable outcome.
  ProQOL questionnaire, scored according to the official ProQOL scoring guidelines. The ProQOL is a validated measure with acceptable internal consistency across its subscales, commonly used to assess compassion fatigue and related constructs in healthcare professionals.
  Descriptive statistics (mean and standard deviation) were calculated. If appropriate, to explore potential sex differences, statistical comparisons were conducted using both Frequentist and Bayesian approaches, with analyses performed in JASP software.

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No